CLINICAL TRIAL: NCT03303261
Title: Study On Discopathie With Modic 1
Status: Terminated | Type: Observational
Why Stopped: The principal investigator decided to stop the study.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: MODIC 1 PRO
Record Dates: First submitted 2017-10-02; First posted 2017-10-06 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2018-03

CONDITIONS: Lumbar Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The chronic lumbago can be associated with an active discopathie, objectified on the MRI by the presence of an inflammatory signal (Modic 1) or greasy (Modic 2) vertebral trays framing the pathological vertebral disk The treatment recommended by t consists in particular of a local infiltration of corticoids which the efficiency is variable according to the patients. The objective of this study is to estimate the efficiency of the local treatment and to highlight some of the factors associated to the advantage of the infiltration by corticoids.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in Rhumatology service for intra-disc infiltration
* Chronic pain (>3 monts)
* VAS >3
* MRI stipulating MODIC 1

Exclusion Criteria:

* radiculalgy
* radicular VAS< lumbar VAS
* pregnancy
* local infection
* corticoid allergy
* previous rachial surgery
* previous spondylodiscite
* psychiatric disorder
* MRI contraindication

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient hospitalized in GHPSJ for infiltration
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
pain VAS ( VISUAL ANALOGIC SCORE) | Day 1 - Day 30

CONTACTS AND LOCATIONS:
Overall Officials: COHEN SOLAL P Julien, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France